CLINICAL TRIAL: NCT02390986
Title: An Extension Study of LON002 in Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LondonPharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LON002-003
Record Dates: First submitted 2015-03-02; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Solid Tumours
Keywords: Cancer; Malignant Neoplasm; Anti-cancer drug
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LON002 — Extension study to provide continuing access to LON002 medication.

SUMMARY:
The purpose of this clinical trial is to evaluate the long term safety and efficacy of LON002.

DETAILED DESCRIPTION:
This is an extension study of LON002 in patients with cancer, who have completed other London Pharma sponsored LON002 studies (parent study). It provides the opportunity for patients to continue receiving treatment for as long as the patient continues to derive a clinical benefit.

Long term safety and efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Has completed a LondonPharma sponsored parent trial of LON002 and continues to have clinical benefit in the judgement of the investigator;
3. Eligible for continuation of LON002 treatment at the end of the parent trial, according to the parent trial protocol;
4. Able to comply with the protocol LON002-003;
5. Women of child bearing potential must have a negative pregnancy test before the start of treatment;
6. Sexually active women of childbearing potential must be using an acceptable form of contraception for the duration of dosing and for 30 days thereafter;
7. Male subjects with female partners of childbearing potential should use condoms for the duration of dosing and for 30 days thereafter

Exclusion Criteria:

1. Has not completed a LondonPharma sponsored parent trial of LON002;
2. Unequivocal evidence of disease progression;
3. Unacceptable toxicity experienced in the parent trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Adverse Events grade ≥3 related to LON002 and Serious Adverse Events related to LON002 as a measure of safety and tolerability. | Participants will be followed for the duration of their study treatment, an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Debashis Sarker, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Mazhar Ajaz, MD, Principal Investigator — Royal Surrey County Hospital NHS Trust; Daryl Bendel, MD, Study Director — Xidea Solutions Ltd
Locations (2):
- United Kingdom (2):
  - The Royal Surrey County Hospital, Guildford, Surrey
  - Guy's and St Thomas NHS Foundation Trust, London